CLINICAL TRIAL: NCT06459323
Title: the Outcomes of Laparoscopic Cholecystectomy for Acute Cholecystitis Within and Beyond the First 72 Hours, Does it Differ?!
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Refaat Mansour, Resident of general surgery Assiut university hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cholecystectomy timing
Record Dates: First submitted 2024-05-15; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Acute Cholecystitis
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic cholecystectomy within first 72hours (Experimental)
  Interventions: Procedure: Laparoscopic cholecystectomy
- Laparoscopic cholecystectomy beyond first 72hours (Experimental)
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Laparoscopic cholecystectomy

SUMMARY:
Compare outcomes of patients undergoing early laparoscopic cholecystectomy within and after72 hours of symptoms.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy (LC) is the mainstay treatment of acute cholecystitis. However, it remains a challenging procedure with low but significant risks of major complications such as bile duct injury increasing as the severity of AC progresses. New Guidelines suggest that laparoscopic cholecystectomy should preferably be performed within 72 hrs of symptom onset but has acknowledged that this may not be always possible in practice. Hence, it recommends that patients presenting after 72 h of symptom onset may still benefit from laparoscopic cholecystectomy in selected patients Studies found that it is imperative to convert to open cholecystectomy when it is deemed unsafe to dissect the Calot's triangle may occur even within or beyond first 72 hrs of attck symptoms. studies found a statistically longer mean total length of hospitalization, operation time and intraoperative blood loss for LC performed beyond 72 h, this did not translate into clinically significant adverse outcomes such as an increase in perioperative morbidity or the need for blood transfusion. After 72 h, chronic inflammation and fibrosis set in resulting in more technically demanding and longer surgeries.Studies show differing results reporting longer operation times for laparoscopic cholecystectomy beyond 72 h, due to stiffer tissues that cannot be bluntly dissected during the subacute phase of tissue inflammation. However, other studies did not report any difference in operation times between both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute cholecystitis within and after 72 hours.
2. Patients over 18 years.
3. Patients with no common bile duct stones based on imaging and biochemical criteria
4. Fit for surgery.

Exclusion Criteria:

1. Patients not fit for surgery
2. Patients with Pancreatitis.
3. Significant medical disease rendering patient unfit for Laparoscopic surgery (e.g. Uncontrolled Diabetes Mellitus, Chronic Pulmonary Disease, significant Cardiac Disease)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Bile duct injury , intraoperative bleeding and operative time | One week
  Evaluate bile duct integrity, calculate amount of blood loss and operative time from the start till the end

REFERENCES:
- See also: Navez, B., Ungureanu, F., Michiels, M. et al. Surgical management of acute cholecystitis: results of a 2-year prospective multicenter survey in Belgium. Surg Endosc 26, 2436-2445 (2012). — http://doi.org/10.1007/s00464-012-2206-7